CLINICAL TRIAL: NCT00737308
Title: Properties and Clinical Performance of Zirconia-based Dental Ceramics
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mahidol University (Other)
Collaborators: Thailand Research Fund (Other)
Responsible Party: Principal Investigator, Kallaya Suputtamongkol, Assistant Professor, Mahidol University
Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MRG5180145
Record Dates: First submitted 2008-08-17; First posted 2008-08-19 (Estimated); Last update posted 2015-05-15 (Estimated); Status verified 2015-05

CONDITIONS: Dental Restoration Wear
Keywords: crowns; ceramics
MeSH Terms: interventions — zirconium oxide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- A (Experimental): crown for clasp
  Interventions: Other: ceramic crown

INTERVENTIONS:
Other: ceramic crown — Zirconia
  Other Names: Zirconia

SUMMARY:
The objectives of this study are to determine the clinical performance of zirconia-based dental prostheses and their related properties.

DETAILED DESCRIPTION:
Zirconia has been used in dentistry since 2000 for constructing fixed partial denture. Its advantages are high fracture resistance, excellent biocompatibility, moderate opacity, etc. Because the increase in demand for more esthetic restoration, zirconia becomes more popular for use as a core material for all-ceramic systems. Its properties have been investigated extensively in many in vitro studies. However, clinical performance of zirconia-based restorations would require a period of time before the results can be assessed. Currently, there are not much results regarding clinical performance of zirconia-based prosthesis and more information are required for future research.

ELIGIBILITY:
Inclusion Criteria:

* Occlusion: At least 20 remaining teeth for each patient, and at least one posterior endodontically treated tooth with natural opposing teeth
* Bruxism: No evidence based on an intraoral exam
* Dental history: No evidence of either moderate or severe periodontal disease
* Medical history: Good to excellent general health

Exclusion Criteria:

* Periodontal status: Pocket depth greater than 4 mm
* Occlusion: Evidence of bruxism or excessive clenching force, Abutment tooth that opposes a removable partial denture, Abutment teeth for fixed partial dentures, Gingival recession of an abutment tooth more than 1 mm from the cementoenamel junction, Tooth with first or second degree of tooth mobility, Tooth with extensive carious lesions

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2008-06; Primary Completion 2015-04 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
ceramic crown fracture | 2 years

SECONDARY OUTCOMES:
masticatory function | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Kallaya Suputtamongkol, Principal Investigator — Mahidol University
Locations (2):
- Thailand (2):
  - Faculty of Dentistry, Mahidol University, Pyathai, Bangkok
  - Faculty of Dentistry, Mahidol University, Bangkok